CLINICAL TRIAL: NCT01763229
Title: The Practical Use of Transthoracic Echocardiography for Obtaining an Optimal Depth of Internal Jugular Venous Catheters in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-1107-116-371
Record Dates: First submitted 2013-01-05; First posted 2013-01-08 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Insertion Depth of Central Venous Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- transthoracic echocardiography (Experimental)
  Interventions: Procedure: transthoracic echocardiography

INTERVENTIONS:
Procedure: transthoracic echocardiography

SUMMARY:
To test if transthoracic echocardiography is useful for correct positioning of central venous catheters in infants with congenital heart disease

DETAILED DESCRIPTION:
Patients scheduled for surgery for congenital heart disease younger than 12 months were studied. Following successful catheter insertion, the insertion depth was determined using transthoracic echocardiography. The long axis or short axis images were used.Chest X-ray images were taken postoperatively and distances from the tip to the carina level were measured.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for surgery under general anesthesia

Exclusion Criteria:

* anomaly of the internal jugular vein
* thrombus in the internal jugular vein

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
the distance between the catheter tip and the carina | After opearation (about 4-6 hour after insertion of the catheter)